CLINICAL TRIAL: NCT03029429
Title: Phase 2 Study of Theophylline Treatment for Pseudohypoparathyroidism
Brief Title: Theophylline Treatment for Pseudohypoparathyroidism
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 133103
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pseudohypoparathyroidism; Albright Hereditary Osteodystrophy
Keywords: pseudohypoparathyroidism; AHO; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Theophylline (Experimental): Theophylline capsules by mouth once daily or Theophylline elixir by mouth q6h (dose determined by serum drug levels)
  Interventions: Drug: Theophylline
- Placebos (Placebo Comparator): Theophylline capsule by mouth once daily or Theophylline elixir by mouth q6h
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Theophylline — oral theophylline
  Other Names: Theo-24, Elixophyllin
  Arms: Theophylline
Drug: Placebos — oral placebo
  Other Names: placebo
  Arms: Placebos

SUMMARY:
Pseudohypoparathyroidism is a genetic disorder with limited treatment options. Patients have early-onset obesity, short stature and increased risk of type 2 diabetes. This phase 2 clinical trial will test the efficacy of theophylline, a phosphodiesterase inhibitor, in pseudohypoparathyroidism. The investigators hypothesize that theophylline will cause weight loss, improve glucose tolerance and slow growth plate closure in children and young adults.

DETAILED DESCRIPTION:
Pseudohypoparathyroidism (PHP) is a rare, genetic disorder caused by impaired stimulatory G protein (Gsα) signaling through downregulation of the gene, GNAS. The resultant hormone abnormalities can be treated with hormone replacement therapy, but other aspects of the disorder such as early-onset obesity and premature epiphyseal closure are without effective treatment options. Gsα signaling is essential for the normal hormonal function of the pituitary, thyroid, gonads, renal proximal tubules and hypothalamus. While many of the resulting hormone deficiencies can be treated with hormone replacement therapy (HRT), HRT is not an effective therapy for the severe early-onset obesity and short stature which are major features of the PHP phenotype. Therefore, the goal of this proposal is to test the efficacy of upstream therapy aimed at correcting the function of two Gsα-dependent receptors responsible for the obesity (melanocortin-4 receptor, MC4R) and short stature (parathyroid hormone, PTH, receptor) phenotype in children with PHP. Gsα-coupled receptor signaling cascade begins with an increase in cyclic adenosine monophosphate (cAMP) which is rapidly degraded by the enzyme phosphodiesterase (PDE). PDE inhibitors act by prolonging cAMP signaling by decreasing the rate of degradation. Given that patients with PHP have reduced, but not completely absent, cAMP production, the investigators seek to test the hypothesis that the PDE inhibitor theophylline will reduce BMI, glucose intolerance, and hormone resistance in children and young adults with PHP through improved Gsα-coupled receptor signaling. The investigators will conduct a 52-week randomized, placebo controlled clinical trial of theophylline in children and young adults with PHP. Theophylline is a non-selective PDE inhibitor that is generically available and has a long history of use in pediatric patients, making it an ideal drug for re-purposing in youth with PHP. Furthermore, the pharmacokinetics of theophylline are well understood and serum drug levels are easily measured. The investigators primary outcome is change in body mass index. Secondary outcome measures include change in glucose tolerance and HRT dose. Anticipating a 10% dropout rate, the investigators will enroll 34 patients and expect that 30 patients will complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13 years and above
2. Clinical diagnosis of PHP (per the EuroPHP network classification guidelines1): Presence of PTH resistance or ectopic classification OR brachydactyly type E plus 2 minor criteria (TSH resistance, other hormonal resistance, developmental delay, intrauterine or post-natal growth retardation, obesity/overweight, specific facial features)
3. Obesity (BMI >95th percentile for age/gender and/or ≥30 kg/m2)

Exclusion Criteria:

1. Use of a PDE inhibitor in the past 30 days
2. History of a seizure disorder unrelated to hypocalcemia
3. History of a cardiac arrhythmia (not including bradycardia)
4. Hepatic insufficiency including cirrhosis and acute hepatitis (AST or ALT >3x upper limit of normal)
5. Congestive heart failure
6. Current cigarette use or alcohol abuse
7. Pregnancy or intention to become pregnant during the next year
8. Untreated hypothyroidism (defined as free thyroxine below the lower limit of normal)
9. Active peptic ulcer disease
10. Current use of medications known to effect theophylline levels
11. History of hypersensitivity to theophylline or other medication components
12. History of Major Depressive Disorder in the past 2 years, lifetime history of suicide attempt, history of any suicidal behavior in the past month, history of other sever psychiatric disorders (e.g. schizophrenia, bipolar disorder)
13. PHQ-9 score is ≥15 or suicidal ideation of type 4 or 5 (C-SSR) in the past month
14. Unable to comply with study procedures in the opinion of the investigator

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | baseline and 52 weeks
  BMI will be expressed a percent of the 95th percentile

SECONDARY OUTCOMES:
Change in insulinogenic index | baseline and 52 weeks
  Insulinogenic index measured during a 75g oral glucose tolerance test
change in levothyroxine dose | baseline and 52 weeks
  levothyroxine dose (mcg/kg/day)
change in calcitriol dose | baseline and 52 weeks
  calcitriol dose (mcg/kg/day)

OTHER OUTCOMES:
Change in body mass index z-score | baseline and 52 weeks
Change in BMI | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Ashley Shoemaker, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoemaker AH, Juppner H. Nonclassic features of pseudohypoparathyroidism type 1A. Curr Opin Endocrinol Diabetes Obes. 2017 Feb;24(1):33-38. doi: 10.1097/MED.0000000000000306. PMID 27875418
- [Background] Wang L, Shoemaker AH. Eating behaviors in obese children with pseudohypoparathyroidism type 1a: a cross-sectional study. Int J Pediatr Endocrinol. 2014;2014(1):21. doi: 10.1186/1687-9856-2014-21. Epub 2014 Oct 15. PMID 25337124
- [Background] Shoemaker AH, Lomenick JP, Saville BR, Wang W, Buchowski MS, Cone RD. Energy expenditure in obese children with pseudohypoparathyroidism type 1a. Int J Obes (Lond). 2013 Aug;37(8):1147-53. doi: 10.1038/ijo.2012.200. Epub 2012 Dec 11. PMID 23229731
- [Background] Mano T, Uchimura K, Hayashi R, Kobahashi T, Fujiwara K, Makino M, Kakizawa H, Nagata M, Nakai A, Wada M, Nagasaka A, Itoh M. Increased urinary phosphate excretion in pseudohypoparathyroidism type II with long-term treatment with phosphodiesterase inhibitor. Horm Metab Res. 1999 Nov;31(11):602-5. doi: 10.1055/s-2007-978804. PMID 10598827
- [Background] Landreth H, Malow BA, Shoemaker AH. Increased Prevalence of Sleep Apnea in Children with Pseudohypoparathyroidism Type 1a. Horm Res Paediatr. 2015;84(1):1-5. doi: 10.1159/000381452. Epub 2015 Apr 23. PMID 25925491
- [Background] Perez KM, Lee EB, Kahanda S, Duis J, Reyes M, Juppner H, Shoemaker AH. Cognitive and behavioral phenotype of children with pseudohypoparathyroidism type 1A. Am J Med Genet A. 2018 Feb;176(2):283-289. doi: 10.1002/ajmg.a.38534. Epub 2017 Nov 28. PMID 29193623
- [Background] Curley KL, Kahanda S, Perez KM, Malow BA, Shoemaker AH. Obstructive Sleep Apnea and Otolaryngologic Manifestations in Children with Pseudohypoparathyroidism. Horm Res Paediatr. 2018;89(3):178-183. doi: 10.1159/000486715. Epub 2018 Feb 16. PMID 29455209
- [Background] Hanna P, Grybek V, Perez de Nanclares G, Tran LC, de Sanctis L, Elli F, Errea J, Francou B, Kamenicky P, Linglart L, Pereda A, Rothenbuhler A, Tessaris D, Thiele S, Usardi A, Shoemaker AH, Kottler ML, Juppner H, Mantovani G, Linglart A. Genetic and Epigenetic Defects at the GNAS Locus Lead to Distinct Patterns of Skeletal Growth but Similar Early-Onset Obesity. J Bone Miner Res. 2018 Aug;33(8):1480-1488. doi: 10.1002/jbmr.3450. Epub 2018 Jun 7. PMID 29693731
- See also: Vanderbilt PHP Research Page — http://www.facebook.com/pseudohypoparathyroidism